CLINICAL TRIAL: NCT02596165
Title: Validation of the Schiller BR-102 Plus PWA Device to Measure Central and Peripheral Hemodynamics
Acronym: BR-102
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopp because of FDA concrns regarding recruitment.
Sponsor: University of Basel (Other)
Collaborators: Kantonsspital Liestal (Other)
Responsible Party: Principal Investigator, Arno Schmidt-Trucksäss, Professor Dr. Arno Schmidt-Trucksäss, University of Basel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EKNZ 2015-327
Record Dates: First submitted 2015-10-28; First posted 2015-11-04 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Aortic Stiffness; Hypertension
Keywords: validation; pulse wave analysis; blood pressure monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pulse wave analysis measurement (Experimental): Measurement of central and peripheral blood pressure and central arterial stiffness simultaneously with the Schiller BR-102 Plus PWA device
  Interventions: Device: Pulse wave analysis measurement with Schiller BR-102 Plus PWA device

INTERVENTIONS:
Device: Pulse wave analysis measurement with Schiller BR-102 Plus PWA device — Measurement of central and peripheral blood pressure and central arterial stiffness simultaneously with the Schiller BR-102 Plus PWA device

SUMMARY:
The significance of parameters of the central hemodynamic is based upon their strong association with left ventricular hypertrophy and target organ damage at the heart. Noninvasive, auscultatory/ oscillometric and therefore easy applicable measurements of the central hemodynamic such as presented by the Schiller BR-102 plus PWA device implicate highly promising potential for research and daily clinical praxis for improved cardiovascular risk assessment on the population level. The purpose of this study is to evaluate the validity of the central and peripheral blood pressure and central arterial stiffness measured with the device BR-102 plus PWA from Schiller (Schiller AG, Baar, Switzerland).

DETAILED DESCRIPTION:
The proposed study is an open, monocentric cross-sectional research study for the evaluation of the validity of the central and peripheral blood pressure and central arterial stiffness measured with the device BR-102 plus PWA from Schiller (Schiller AG, Baar, Switzerland). For that purpose measurement of the respective parameters in cardiovascular disease free individuals will be compared with validated devices and the agreement between the devices will be statistically analyzed. Central blood pressure and central arterial stiffness are clinically increasingly meaningful parameters of the cardiovascular system that allow improved, early cardiovascular risk stratification. The significance of parameters of the central hemodynamic is based upon their strong association with left ventricular hypertrophy and target organ damage at the heart. Noninvasive, auscultatory/ oscillometric and therefore easy applicable measurements of the central hemodynamic such as presented by the Schiller BR-102 plus PWA device implicate highly promising potential for research and daily clinical praxis for improved cardiovascular risk assessment on the population level.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals free of clinically relevant cardiovascular diseases or diabetes based on medical history and physical examination.
* Heart rhythm: Sinus rhythm
* Blood pressure range: 10 to 12 subjects in each of the three systolic blood pressure (SBP) and three diastolic blood pressure (DBP) recruitment ranges (low, medium, high).

Exclusion Criteria:

* Cardiac arrhythmia (atrial fibrillation, frequent extrasystoles)
* Pacemaker-dependent
* Pregnancy after the 6th month of the pregnancy
* Body mass index (BMI)>30 kg/m2
* Known significant carotid or femoral artery stenosis
* Impalpable arterial pulse at site of measurement
* Age under 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
central blood pressure | 1 day
  Measurement of central blood pressure and central arterial stiffness simultaneously with the Schiller BR-102 Plus PWA device
central arterial stiffness | 1 day
  Measurement of central blood pressure and central arterial stiffness simultaneously with the Schiller BR-102 Plus PWA device

SECONDARY OUTCOMES:
peripheral blood pressure | 1 day
  Measurement peripheral blood pressure with the Schiller BR-102 Plus PWA device

CONTACTS AND LOCATIONS:
Overall Officials: Arno Schmidt-Trucksäss, MD, MA, Principal Investigator — Department for Sport, Exercise and Health, Sports and Exercise Medicine, University of Basel, Basel, Switzerland, 4052